CLINICAL TRIAL: NCT01315184
Title: Pilot Trial of a Therapeutic Interactive Voice Response System for Buprenorphine Maintenance: The Recovery Line Support System
Brief Title: Study of Computer-Based Treatment for Drug Dependence
Acronym: RLSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0804003684; K01DA022398-01A2 (NIH)
Record Dates: First submitted 2010-09-16; First posted 2011-03-15 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Opioid-Related Disorders; Heroin Dependence
Keywords: Interactive Voice Response; Computer-based Treatment; Opioid Agonist; Buprenorphine; Methadone
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recovery Line Support System (Experimental): Patients assigned to the Recovery Line Support System will be trained on the system and provided 24-hr access to the system for a four week period, provided with a Recovery notebook, and given reminder calls to contact the system.
  Interventions: Behavioral: Recovery Line Support System
- Treatment as Usual (No Intervention): Patients assigned to the TAU condition will receive any services provided by their buprenorphine provider and any additional services that their provider refers or recommends that patients attend. No additional services will be provided by the study.

INTERVENTIONS:
Behavioral: Recovery Line Support System — Full time access (24 hours/7 days per week) to an automated, telephone-based, interactive, voice response (IVR)system for 4 weeks.
  The program was developed based on a behavioral theory of substance abuse, and comprises four components: 1) self-assessment 2) learning about skills , 3) activities for current help and skills training, and 4) Feedback.
  Arms: Recovery Line Support System

SUMMARY:
The purpose of this study is to evaluate the whether an automated telephone-based system is useful and helpful for opioid dependent patients receiving buprenorphine in primary care. The Recovery Line support system is a Therapeutic Interactive Voice Response system based on cognitive behavioral therapy (CBT). The Recovery Line support system includes a variety of modules presenting the basic principles and strategies of CBT. Each module includes learning sections and activities sections to provide direct guidance in using skills. The Recovery Line support system is interactive and also includes a questionnaire to help patients identify problems and recommend modules for use, as well as an inspiration section, an introduction, and an immediate assistance menu. Following development of an initial system the current trial will recruit 40 patients receiving buprenorphine maintenance from a physician provider in the local community. Patients will be randomly (flip of a coin) to receive the Recover Line Support system or to treatment as usual with their physician. Patients assigned to TIVR will be trained on the system and provided 24-hr access to the TIVR system for a four week period. Primary outcome variables will be how long patients remain in treatment, self-reported abstinence from opioids and other drugs, and abstinence as measured by weekly drug screens. It is expected that patients assigned to TIVR will better treatment outcomes than patients assigned to TAU.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years old
* have initiated buprenorphine maintenance treatment from an approved physician in the previous two weeks

Exclusion Criteria:

* are a current suicide or homicide risk or meet criteria for psychiatric disorder that would interfere with ability to complete study
* are unable to read or understand English
* have a life-threatening or unstable medical problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Opioid Abstinence | 4 Weeks
  Continuous opioid abstinence as documented by weekly urinalysis
Retention | 4 Weeks
  Retention in the study

SECONDARY OUTCOMES:
Self Reported Drug Abstinent | 4 weeks
  Drug Abstinence based on weekly interviews
system use | 4 weeks
  Call total amount, frequency, and specific system utilization

CONTACTS AND LOCATIONS:
Overall Officials: Brent A. Moore, Ph.D., Principal Investigator — Yale University
Locations (1):
- APT Foundation, New Haven, Connecticut, United States